CLINICAL TRIAL: NCT04298866
Title: White Matter Hyperintensities Subtypes in Cerebral Small Vessel Disease : 7 Tesla Ultra-high Resolution Imaging MRI
Acronym: SV7
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180445
Record Dates: First submitted 2020-02-26; First posted 2020-03-06 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Other)
  Interventions: Other: Experimental Arm

INTERVENTIONS:
Other: Experimental Arm — * 3T MRI, maximum 1H30 long duration, including diffusion tensor imaging, susceptibility weighted imaging, multiparametric acquisitions, without contrast perfusion acquisitions.
  * 7T MRI, maximum 1H30 long duration, including contrast enhanced acquisitions
  * Neuropsychological battery including chronometric measures obtained through a computer interface

SUMMARY:
Cerebral small vessel diseases (SVD) are a very frequent group of disorders all characterized by alterations of the structure and/or function of small arteries, veins and capillaries. In these disorders, brain tissue lesions accumulate years before the occurrence of clinical symptoms which can be devastating such as stroke, cognitive disturbances and gait disorders. So far, chronic hypoperfusion was considered to be responsible for the accumulation of such lesions. However, recent results have suggested that the lesions underlying white matter hyperintensities (WMH), the most common MRI marker of SVD visible on conventional MRI in quite every subject with SVD long before the occurrence of clinical events, may depend on the considered brain area and may correspond to various mechanisms. Some WMH may even be associated with less severe clinical manifestations.The aim of the present study is to identify different types of WMH by studying 100 patients with different forms of SVD with the most advanced MRI (including ultra-high-resolution imaging at 7 Tesla, new diffusion protocol, sodium MRI, contrast-enhanced angiography and relaxometry and post-processing techniques), and post-processing techniques (machine learning, deep learning, artificial intelligence).

ELIGIBILITY:
Inclusion Criteria:

* Subjects or patients with MRI defined cerebral small vessel disease including different extents of white matter hyperintensities, presumably related to hypertension (30 patients), cerebral amyloid angiopathy (30 patients), CADASIL (30 patients) or any other monogenic form of cerebral small vessel disease (HTRA1 AD, COLIVA1… 10 patients)
* Age ≥ 18 years
* No dementia (MMSE > 24 and absence of dependence in daily activities)
* No disability (modified Rankin's scale < 2)
* No history of severe allergic reaction, in particular to gadolinium infusion
* No history of severe asthma
* No renal insufficiency (clearance < 60 ml/mn/1.73 m2)

Exclusion Criteria:

* Contraindications to MRI
* Standard MRI of bad quality due to movement artefacts
* Dementia or disability
* Patient without affiliation to the French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-06-04 (Estimated); Study Completion 2023-06-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a different form of white matter hyperintensities (WMH) | at the time of specific imaging (between Day 1 to Day 60)
  The different forms of white matter hyperintensities will be assessed and identified using MRI imaging.The pattern of co-variation of structural, functional, metabolic imaging modalities, estimated in each voxel of a reference space, both inside and outside the WMH, will be compared through massive statistical approaches, controlled, for multiple testing

SECONDARY OUTCOMES:
Frequency of different WMH subtypes in different types of small cerebral vessel disease | at the time of specific imaging (between Day 1 to Day 60)
  Distribution of white matter hyperintensities in different brain areas according to the small cerebral vessel disease
Frequency of large tract involvement | at the time of specific imaging (between Day 1 to Day 60)
  Large tratreconstructed from diffusion imaging) by WMH depending on the the small cerebral vessel disease
Global cognitive function | at inclusion
  The global cognitive functions will be assessed using MOCA. The MoCA assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation to time and place
Language | at inclusion
  Language assessment will be done using LAST and Boston Naming Test
Spatial exploration | at inclusion
  The neglect and spatial exploration will be assessed with bells test from the BEN neglect battery
Spatial memory | at inclusion
  Spatial memory will be assessed using the brief visual-spatial memory test (BVMT-R)
Visual memory | at inclusion
  Visual memory will be assessed using the brief visual-spatial memory test (BVMT-R)
Episodic verbal memory | at inclusion
  Episodic verbal memory test by the RL RI 16
Working memory | at inclusion
  Working memory will be evaluated by the working memory index of the WAIS-IV
Executive function | at inclusion
  Executive function will be assessed by the versions A and B of the Trail Making Test
Attentional Performances status | at inclusion
  Attentional Performances will be assessed using a battery on a computer which tests different attentionnal and executive function
Depression and Anxiety status | at inclusion
  Depression and anxiety will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire. The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Apathy status | at inclusion
  Apathy status will be assessed using the Starkstein scale
Pulse wave Velocity count | at inclusion
  Arterial stifness will be assessed by measuring the pulse wave velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lariboisière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided